CLINICAL TRIAL: NCT02137863
Title: Phase 4 Study of Dexmedetomidine Effects on Preventing Contrast Induced Nephropathy
Brief Title: Efficacy of Dexmedetomidine in Preventing Contrast Induced Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Aynur Akın, Prof Dr, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011/345
Record Dates: First submitted 2014-01-13; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: Contrast induced nephropathy; Diabetes Mellitus; Dexmedetomidine
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Before the angiography 0.9 % sodium chloride 3 ml/kg/h administered for 12 hours.
  During the angiography and 12 hours after angiography 1 ml/kg/h 0.9 % sodium chloride administered.
  100 ml/10min 0.9 % NaCl administered intravenously just before the angiography.
  1 ml/kg/h 0.9 % sodium chloride administered intravenously during the procedure and was continued 1 hour after the angiography.
  Interventions: Drug: 0.9 % NaCl
- Dexmedetomidine (Active Comparator): Before the angiography 0.9 % sodium chloride 3 ml/kg/h administered for 12 hours.
  During the angiography and 12 hours after angiography 1 ml/kg/h 0.9 % sodium chloride administered.
  Dexmedetomidine was diluted as 1 μg/ml. 1 μg/kg/10min dexmedetomidine administered intravenously just before the angiography.
  1 μg/kg/h dexmedetomidine administered intravenously during the procedure and was continued 1 hour after the angiography.
  Interventions: Drug: Dexmedetomidine; Drug: 0.9 % NaCl

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenously 1μg/kg/10min administered just before the procedure.
  1 μg/kg/h administered during the angiography and was continued 1 hour after the angiography.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: 0.9 % NaCl — During 12 hours before the procedure 3 ml/kg/h 0.9 % NaCl infusion and 1 ml/kg/h during the angioplasty and 12 hours after the procedure.
  Other Names: Normal Saline
Drug: 0.9 % NaCl — 100 ml/10min infusion just before the angiography
  1 ml/kg/h infusion during the angiography and was continued 12 hours after the procedure
  Other Names: Normal Saline
  Arms: Control

SUMMARY:
The aim of this study was to evaluate the effects of dexmedetomidine on renal function, hormonal and hemodynamic parameters in contrast media induced diabetic patients.

DETAILED DESCRIPTION:
Contrast nephropathy may occur after using intravenous contrast media and may result in acute renal failure. Contrast nephropathy usually reversible but in some cases it can be permanent. This situation increase the time of hospitalization and mortality of the patients. Although the only proved prevention from contrast nephropathy method is hydration, infusion of dexmedetomidine may keep the renal functions.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for percutaneous coronary angiography
* > 18 yo
* Diabetic patients
* Creatinin value < 3 mg/dl

Exclusion Criteria:

* Contrast agent hypersensitivity
* Pregnant patients
* Creatinin value ≥3mg/dl
* patients have acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes in glomerular renal function after percutaneous coronary angiography as measured by neutrophil gelatinase-associated lipocalin, cystatin c, blood urea nitrogen, creatinin | 1 day (from start of angioplasty till discharge from the hospital)

SECONDARY OUTCOMES:
blood pressure | 1 day (from start of angiography till discharge from the hospital)
Heart rate | 1 day (from start of angiography till discharge from the hospital)
Blood electrolyte levels ( sodium, potassium, chloride) | before the angiography and just before the discharge from hospital
complete blood count | before the angiography and just before the discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Akın, Prof, Study Chair — TC Erciyes University